CLINICAL TRIAL: NCT07388914
Title: Aldosterone Variations in Patients With Primary Hyperparathyroidism Before Surgery and in the Year Following Surgery for Parathyroid Disease.
Brief Title: Aldosterone Variations in Patients With Primary Hyperparathyroidism After Surgery
Acronym: ALDOPARA2
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, NOMINE-CRIQUI Claire, MD-Head of the endocrine surgery Unit, Central Hospital, Nancy, France
Other Study IDs: 2026PI016
Record Dates: First submitted 2026-01-27; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Primary Hyperparathyroidism; Primary Hyperparathyroidism Due to Adenoma
Keywords: aldosteron; primary hyperparathyrodism; hypertension
MeSH Terms: conditions — Hyperparathyroidism, Primary; Parathyroid Neoplasms; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with primary hyperparathyroidism: Patients with primary hyperparathyroidism who are candidates for surgery. All patients underwent biological testing for parathyroid hormone, calcium, aldosterone, renin and renal function.
  Their blood pressure was measured five times during the pre-operative consultation and after surgery.
  Their antihypertensive treatments were collected prior to surgery and after.

SUMMARY:
Primary hyperparathyroidism is a disorder of calcium and phosphorus metabolism linked to dysfunction of one or more parathyroid glands. The latest recommendations from the American Association of Endocrine Surgeons (7) consider the presence of hypertension as an argument for proposing the removal of a parathyroid adenoma in the context of primary hyperparathyroidism. The renin-angiotensin-aldosterone system is involved in regulating blood pressure.

The main objective of this study is to assess aldosterone level in patients with primary hyperparathyroidism before surgery and its variation in the year following surgery for parathyroid disease.

Secondary objectives are to assess aldosterone variations after surgery at 3 months

* Assess aldosterone variations after surgery at 6 months
* Assess aldosterone variations after surgery at 12 months
* Blood pressure changes before and after surgery (5 pre- and post-operative measurements)
* Assess the number of antihypertensive treatments before and after surgery
* Assess antihypertensive treatment according to the WHO-DDD classification before and after surgery Compare aldosterone levels in the 'primary hyperparathyroidism' group with a control group of patients from the general population (using the STANISLAS cohort).

  * Compare aldosterone levels in the HPT group with aldosterone levels in a group of patients after myocardial infarction (cardiovascular patient group )

DETAILED DESCRIPTION:
Primary hyperparathyroidism is a disorder of calcium and phosphorus metabolism linked to dysfunction of one or more parathyroid glands, without any underlying chronic kidney disease. The disease manifests itself in its classic forms as elevated blood calcium, parathyroid hormone and calcium levels. It has an impact on bone mineralisation, the presence of kidney stones, glucose metabolism (1)(2) and cardiovascular function (3)(4)(5).

A Scottish study published in 2023, based on a robust medical information system enabling prospective follow-up, showed an overall prevalence of primary hyperparathyroidism between 2007 and 2018 of 0.84%, which was much higher in women (1.18%) than in men (0.48%) (6) The latest recommendations from the American Association of Endocrine Surgeons (7) consider the presence of hypertension as an argument for proposing the removal of a parathyroid adenoma in the context of primary hyperparathyroidism: 'Parathyroidectomy may be offered to surgical candidates with cardiovascular disease who might benefit from mitigation of potential cardiovascular sequelae other than hypertension.' There appears to be an association between hypertension and primary hyperparathyroidism (4)(5). Its mechanism is currently poorly understood and little described. Using the keywords 'hyperaldosteronism' AND 'hyperparathyroidism', we found only one case report (in Spanish) and one article, but these focused more on patients already suffering from primary hyperaldosteronism (8)(9).

The renin-angiotensin-aldosterone system is involved in regulating blood pressure.

This is why we systematically measure aldosterone and renin preoperatively and at three postoperative points following surgery for primary hyperparathyroidism.

This is a retrospective study including among 400 patients with primary hyperparathyroidism. Allt his patients underwent parathyroidectomy.

Inclusion critera : patients with primary hyperparathyroidism, age>18 years Exclusion criteria : patients with hyperparathyroidism and renal insuffisency Pregant women, patients < 18 years. All patients underwent blood tests including PTH, calcium, aldosterone and renin levels before surgery and 3 months, 6 months and 12 months after surgery.

The number and type of antihypertensive treatments were systematically recorded before and 3 months after surgery.

In a second step, the aldosterone levels of patients with primary hyperparathyroidism will be compared with a cohort of patients from the general population: the STNISLAS cohort, and with a cohort of patients with cardiovascular disease. This will enable to identify whether aldosterone levels in the population of patients with primary hyperparathyroidism differ from those in the general population.

The Main objective is to assess the role of phosphorus-calcium metabolism on the renin-angiotensin system in patients with primary hyperparathyroidism (PHPT)

The Secondary objectives are :

1. To describe the evolution of the renin-angiotensin system (plasma aldosterone and renin levels) before and after parathyroidectomy (at 3, 6 and 12 months) in patients with PHPT.
2. To evaluate the links between changes in phosphorus-calcium metabolism and variations in plasma aldosterone and renin levels after surgery for PHPT.
3. To evaluate changes in the number and dosage (WHO-DDD classification) of antihypertensive medications before and after surgery for PHPT.
4. To evaluate changes in blood pressure values before and after surgery for PHPT (five measurements).
5. To evaluate the links between blood pressure values before and after surgery for PHPT and changes in plasma aldosterone and renin levels.
6. To compare the renin-angiotensin system (plasma aldosterone and renin levels) in patients with PHPT versus healthy patients from the general population (STANISLAS cohort)

8) To compare the renin-angiotensin system (plasma aldosterone and renin levels) in patients with PHPT versus patients with cardiovascular disease (REMI cohort)

ELIGIBILITY:
Inclusion Criteria:

* patients with primary hyperparathyroidism candidate to surgery
* age>/=18 years

Exclusion Criteria:

age< 18 years patients with renal insufficiency (CKDEpi <60ml/mn) pregant women

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary hyperparathyroidism, without renal insufficiency , candidate to parathyroid surgery
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Aldosteron variation before and after surgery | from enrollment to 12 months after surgery
  Variation of aldosteron level between the time before surgery and after surgery at 3 points : 3,6 and 12 months after surgery

SECONDARY OUTCOMES:
Plasma Parathormon levels | 3 months before surgery to 12 months after surgery The measure is done at 3,6 and 12 months after surgery
  Preoperative and postoperative Plasma parathormone levels
Plasma Calcium and Phosphorus levels | 3 months before surgery to 12 months after surgery The measure is done at 3,6 and 12 months after surgery
  Preoperative and postoperative Plasma calcium and phosphorus levels
Plasma renin levels | 3 months before surgery to 12 months after surgery The measure is done at 3,6 and 12 months after surgery
  Preoperative and postoperative Plasma renin levels
type and number of antihypertensive medications | from 3 months before surgery to 3 months after
  Preoperative and postoperative type and number of antihypertensive medications : the number, the type and the dosage of anti-hypertensive drugs is collected before and 3 months after surgery
WHO_DDD classification | from 3 months before surgery to 3 months after
  Using the WHO_DDD classification , a score of anti-hypertensive medication is calculated before and after surgery for each patient.
Systolic and diastolic blood pressure (SBP and DBP) | from 3 months before surgery to 3 months after
  Preoperative and postoperative SBP and DBP value in mmHg are systematically measured 3 months before and 3 months after surgery.
Preoperative glomerular filtration rate (GFR) | 3 months before surgery.
  Preoperative glomerular filtration rate (GFR) is measured before surgery. Patients with renal insufficiency are excluded.
Preoperative 25 OH vitD | 3 months before surgery
  Plasma of 25OH vitamin D before surgery
Preoperative 24h calciuria | 3 months before surgery
  24h calciuria 3 months before surgery
Kidney stones | 3 months before surgery
  Presence of kidney stones on ultrasound or abdominal CT scan prior to parathyroid surgery
femoral T score | 3 months before surgery
  Femoral T-score on preoperative bone densitometry

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nancy, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martin Navarro JA, Medina Zahonero L, Procaccini FL, Barba Teba R, Rubio Menendez V, Valle Alvarez E, PoloCanovas ME, Ortega-Diaz M, Puerta Carretero M, Lucena Valverde R, Munoz Ramos P, Alcazar Arroyo R, de Sequera Ortiz P. Hyperaldosteronism and hyperparathyroidism. A disturbing friendship. Nefrologia (Engl Ed). 2024 Jul-Aug;44(4):496-502. doi: 10.1016/j.nefroe.2024.07.007. Epub 2024 Aug 5. PMID 39107222
- [Background] Araujo-Castro M, Pascual-Corrales E, Fernandez-Argueso M, Bengoa-Rojano N, Garcia Cano A, Jimenez Mendiguchia L, Cuesta M. The prevalence of primary and secondary hyperparathyroidism and its cardiometabolic implications in primary aldosteronism. Minerva Endocrinol (Torino). 2023 Dec;48(4):401-410. doi: 10.23736/S2724-6507.23.03866-6. Epub 2023 May 11. PMID 37166400
- [Background] Wilhelm SM, Wang TS, Ruan DT, Lee JA, Asa SL, Duh QY, Doherty GM, Herrera MF, Pasieka JL, Perrier ND, Silverberg SJ, Solorzano CC, Sturgeon C, Tublin ME, Udelsman R, Carty SE. The American Association of Endocrine Surgeons Guidelines for Definitive Management of Primary Hyperparathyroidism. JAMA Surg. 2016 Oct 1;151(10):959-968. doi: 10.1001/jamasurg.2016.2310. PMID 27532368
- [Background] Soto-Pedre E, Newey PJ, Leese GP. Stable Incidence and Increasing Prevalence of Primary Hyperparathyroidism in a Population-based Study in Scotland. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e1117-e1124. doi: 10.1210/clinem/dgad201. PMID 37022975
- [Background] Kalla A, Krishnamoorthy P, Gopalakrishnan A, Garg J, Patel NC, Figueredo VM. Primary hyperparathyroidism predicts hypertension: Results from the National Inpatient Sample. Int J Cardiol. 2017 Jan 15;227:335-337. doi: 10.1016/j.ijcard.2016.11.080. Epub 2016 Nov 9. PMID 27847154
- [Background] Han D, Trooskin S, Wang X. Prevalence of cardiovascular risk factors in male and female patients with primary hyperparathyroidism. J Endocrinol Invest. 2012 Jun;35(6):548-52. doi: 10.3275/7861. Epub 2011 Jul 12. PMID 21750400
- [Background] Al-Jehani A, Al-Ahmed F, Nguyen-Thi PL, Bihain F, Nomine-Criqui C, Demarquet L, Guerci B, Ziegler O, Brunaud L. Insulin resistance is more severe in patients with primary hyperparathyroidism. Surgery. 2022 Aug;172(2):552-558. doi: 10.1016/j.surg.2022.02.012. Epub 2022 Apr 1. PMID 35379519
- [Background] Koubaity O, Mandry D, Nguyen-Thi PL, Bihain F, Nomine-Criqui C, Demarquet L, Croise-Laurent V, Brunaud L. Coronary artery disease is more severe in patients with primary hyperparathyroidism. Surgery. 2020 Jan;167(1):149-154. doi: 10.1016/j.surg.2019.05.094. Epub 2019 Oct 24. PMID 31668778
- [Background] Nomine-Criqui C, Bihain F, Nguyen-Thi PL, Scheyer N, Demarquet L, Klein M, Guerci B, Brunaud L. Patients with prediabetes improve insulin resistance after surgery for primary hyperparathyroidism. Surgery. 2024 Jan;175(1):180-186. doi: 10.1016/j.surg.2023.04.072. Epub 2023 Nov 18. PMID 37981555